CLINICAL TRIAL: NCT05922358
Title: Observation of Oxaliplatin Hypersensitivity and Neurotoxicity in GI Tract, and Reuse of Oxaliplatin Hypersensitivity in Gastrointestinal Tumors: A Prospective, Open-Label, Multicenter, Phase II Study
Brief Title: Phase II Study of Reuse of Oxaliplatin Hypersensitivity in Gastrointestinal Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-027
Record Dates: First submitted 2023-06-18; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Gastrointestinal Tumors
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypersensitivity group (Experimental): Corresponding intervention measures are given for different levels of hypersensitivity reactions
  Interventions: Combination Product: Anti-allergic treatment

INTERVENTIONS:
Combination Product: Anti-allergic treatment — For grade I-III hypersensitivity to oxaliplatin, oxa 0.01 mg/ml, 0.1 mg/ml and 5 mg/ml were used in sequence for skin test. 5% GS was used as a negative control. Test results are read within 15 to 20 minutes.
  Grade IV: Permanently stop using oxaliplatin; Grade I-II: Take orally (cetirizine 10 mg bid, dexamethasone 8 mg bid, ranitidine 150 mg bid*3dose) the day before the next cycle of oxaliplatin. The infusion rate is 50% of the original rate; if a grade II hypersensitivity reaction occurs again, the treatment method is the same as that of a grade III hypersensitivity reaction.
  Grade III: Oral drugs are the same as above. 0.5h before oxaliplatin: dexamethasone 10mg iv, cimetidine 40mg iv, promethazine 25mg im. The first bag of 10% total amount of oxaliplatin + 5% GS500ml: 5ml/h*1h, 45ml/h*1h, then 225ml/h*2 hours; then dexamethasone 10mg iv; the second bag of 90% total Oxa +5%GS500ml: 100ml/h*0.5h, then 150ml/h*3 hours.

SUMMARY:
The incidence of oxaliplatin allergy reactions is between 12-15%, while the incidence of severe (grade 3-4) allergic reactions is between 0.5-2%. The purpose of this study is to prospectively investigate the incidence of oxaliplatin allergy and neurotoxicity, and to evaluate the use of effective anti-allergic and desensitization therapies to enable patients who are already allergic to oxaliplatin to complete their prescribed doses smoothly.

DETAILED DESCRIPTION:
The incidence of oxaliplatin allergy reactions is between 12-15%, while the incidence of severe (grade 3-4) allergic reactions is between 0.5-2%. The purpose of this study is to prospectively investigate the incidence of oxaliplatin allergy and neurotoxicity, and to evaluate the use of effective anti-allergic and desensitization therapies to enable patients who are already allergic to oxaliplatin to complete their prescribed doses smoothly.

Patients with GI receiving oxaliplatin-containing regimens were prospectively observed, and patients with oxaliplatin grade I-III hypersensitivity reactions judged by clinicians based on clinical symptoms and signs entered the oxaliplatin reuse study . For patients with grade I-III oxaliplatin allergy, oxaliplatin skin test with 3 concentration gradients (0.01 mg/ml, 0.1 mg/ml and 5 mg/ml) was performed, and 5% glucose Water served as a negative control. 15-20 minutes to read test results. If the largest diameter of the rash was greater than 3 mm of the negative control, it was judged as a positive result. Afterwards, interventions were performed in different ways according to the grade of oxaliplatin allergic reaction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who plan to receive oxaliplatin treatment;
2. Male or female aged 18-75 year;
3. ECOG PS 0-2;
4. The expected survival time is more than 3 months;
5. Capable and willing to accept survey patients

Exclusion Criteria:

1.Patients who were not suitable for the enrollment of this study judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Completion rate of 3 cycles of re-chemotherapy with oxaliplatin | 2 years
  Completion rate of 3 cycles of re-chemotherapy with oxaliplatin

SECONDARY OUTCOMES:
Concordance rate between oxaliplatin skin test results and clinicians' judgment | 2 years
  Concordance rate between oxaliplatin skin test results and clinicians' judgment